CLINICAL TRIAL: NCT05838287
Title: Pioglitazone, Lipotoxicity, and Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Pioglitazone on Heart Failure in Type-2 Diabetes Mellitus Participants
Acronym: PIOHF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20220916H
Record Dates: First submitted 2023-04-10; First posted 2023-05-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: double-blind placebo controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the participant nor the investigator knows what treatment is given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pioglitazone Administration Group (Active Comparator): Pioglitazone 15mg/day titrated to 30 mg/day at week 2 and to 45 mg/day at week 4
  Interventions: Drug: Pioglitazone
- Placebo/Control Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Participants will be taking Pioglitazone tablets 1/day for 24 weeks.
  Other Names: Actos
  Arms: Pioglitazone Administration Group
Drug: Placebo — Placebo for Pioglitazone
  Other Names: Placebo tablet
  Arms: Placebo/Control Group

SUMMARY:
Our goal of the study is to learn the effects of the diabetes medication named Pioglitazone, in type-2 diabetic obese participants with Heart failure. The main question it aims to answer are:

1. To demonstrate that impaired mitochondrial function leading to reduced ATP generation plays a key pathophysiologic role in the development of heart failure with preserved ejection fraction (HFpEF) in obese type 2 diabetic (T2D) individuals.
2. To demonstrate that pioglitazone, improves diastolic (as well as systolic) function by improving myocardial insulin sensitivity and by reducing both myocardial and epicardial fat content.

DETAILED DESCRIPTION:
Either Pioglitazone or Placebo Pioglitazone will be administered during this study in this Type 2 Diabetic population with Heart Failure to examine if there are any beneficial effects on diastolic and systolic function.

Myocardial blood flow (MBF) is measured using a PET scan, then participants will be randomized to pioglitazone or a placebo to examine the effects of the study drug on the effects on the systolic and diastolic function of the heart. In addition, myocardial insulin sensitivity change will be measured as well as myocardial fat content. The ratio of ATP: PCr will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 30-70 years
4. Body Mass Index (BMI) of 27.5-40kg/m²
5. HbA1c of 6.5 to 10%
6. Blood pressure of less than or equal to 145/65mmHg
7. eGFR greater than 45 ml/min/1.73m²
8. Subject must have HFpEF (EF > 50% by ECHO screening)
9. NYHA class II-III heart failure
10. Only T2D patients treated with diet/exercise, metformin, sulfonylurea, metformin/SU, DPP4i or insulin will be studied.
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional [4 weeks] after the end of study participation.
12. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Subjects with history of osteoporosis or proliferative diabetic retinopathy
2. Subjects with Heart failure due to restrictive or infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, severe valvular heart disease, etc. will be excluded
3. Patients with symptomatic coronary artery disease.
4. Subjects with significant change in diuretic management during the month prior to screening (defined by doubling of diuretic dose, or addition of another HF medication).
5. Subjects treated with a GLP-1 RA or thiazolidinedione.
6. Subjects treated with a SGLT2i
7. Pregnancy or lactation
8. Known allergic reactions to components of the study interventions.
9. Any metal plates, parts, screws, shrapnel, pins in body, or cardiac (heart) pacemaker

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic function | Baseline and 6-months post treatment (approximately 24 weeks)
  Measurement of change in systolic function of the heart using cardiac MRI
Change in Diastolic function | Baseline and 6-months post treatment (approximately 24 weeks)
  Measurement of change in diastolic function of the heart using cardiac MRI

SECONDARY OUTCOMES:
Myocardial insulin sensitivity | Baseline and 6-months post treatment (approximately 24 weeks)
  Measurement of change in Free Plasma Glucose (FPG) in blood plasma
Myocardial fat content | Baseline and 6-months post treatment (approximately 24 weeks)
  Measurement of change in myocardial fat content
PCr:ATP ratio | Baseline and 6-months post treatment (approximately 24 weeks)
  Measurement of change in PCr:ATP ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — University of Texas
Locations (1):
- Texas Diabetes Institute/UH, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be available to other researchers.